CLINICAL TRIAL: NCT02135601
Title: The Effects of the Water-exchanged Colonoscopy on Adenoma Detection Rate: a Multicenter, Randomized, Single Blind, Control Trial
Brief Title: The Effects of the Water-exchanged Colonoscopy on Adenoma Detection Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20140408-7
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-08

CONDITIONS: Adenoma; Pain
Keywords: colonoscopy; water; adenoma; pain
MeSH Terms: conditions — Adenoma; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air colonoscopy (No Intervention): Colonoscopy will be performed without medications and with judicious air insufflation during colonoscope insertion.
- Water colonoscopy (Other): Colonoscopy will be performed without medications and aided by water infusion in-lieu of air insufflation during insertion of the colonoscope.
  Interventions: Other: Water colonoscopy

INTERVENTIONS:
Other: Water colonoscopy — Colonoscopy will be performed without medications and aided by water infusion in-lieu of air insufflation during insertion of the colonoscope. The water infusion involves putting warm sterile water into the colon to open up the colon for advancement of the colonoscope until the end of the colon (cecum) is reached. The water is delivered through scope irrigation channel by an infusion pump equipped with a foot switch which will be controlled by the endoscopist. Infused water used to cleanse residual fecal matter will be suctioned as needed to clear the colonic lumen.
  Arms: Water colonoscopy

SUMMARY:
Water exchange method has been shown to reduce medication requirement and pain experienced during colonoscopy. It may increase the adenoma detection rate (ADR). Water exchange provides salvage cleansing and the refractive index of water (n equals about 1.3) is larger than that of air, which creates optical distortion that likely contributes to objects appearing larger underwater, making smaller lesions easier to visualize and it may help draw attention to those smaller lesions during withdraw. These principles facilitate to the higher adenoma detection rate.

There is a large number of literature on the adenoma detection rate during water exchange colonoscopy, but most studies have been conducted in only one centre, simple-size, and under sedation patients, the influence of adenoma detection rate under unsedation patients was unclear.

The aim of this study is to compare the ADR of colonoscopy by using the water exchange method versus the conventional air method in unsedation patients in multiple centers in China.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 patients with intact colon and rectum

Exclusion Criteria:

* prior finding of severe colorectal stricture;
* solid fetus contained in the last stool before colonoscopy
* no bowel preparation or cleansed by enema/lavage
* without the requirement of reaching cecum
* known colorectal polyps or polyposis syndrome without complete removal previously
* pregnant women
* hemodynamically unstable
* patients who cannot give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3303 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | up to one year
  The proportion of participants with at least one adenoma in each group

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | up to one year
  0 = no pain, to 10 = most severe pain
Cecal intubation success rate | up to one year
  Insertion of a colonoscope to the cecum
Cecum intubation time | up to one year
  Total time of colonoscope intubation from anus to cecum
Quality of Bowel Preparation | up to one year
  BBPS：cleanliness of each part of the colon: 0=unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared; 1=portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen because of staining, residual stool, and/or opaque liquid; 2=minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well; 3=entire mucosa of colon segment seen well with no residual staining, small frag- ments of stool, or opaque liquid.

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Principal Investigator — Air Force Military Medical University, China; Felix W. Leung, M.D., Principal Investigator — Sepulveda Ambulatory Care Center, VAGLAHS
Locations (6):
- China (6):
  - Chaoyang Hospital, Beijing, Beijing Municipality
  - General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - Union Hospital of Tongji Medical college, Wuhan, Hubei
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Renji Hospital, Shanghai, Shanghai Municipality
  - First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang